CLINICAL TRIAL: NCT00290095
Title: Quality of Life in Patients With Multiple Myeloma
Status: Completed | Type: Observational
Sponsor: Ullevaal University Hospital (Other)
Organization: Oslo University Hospital (Other)
Other Study IDs: 1.2005.1269
Record Dates: First submitted 2006-02-09; First posted 2006-02-10 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2011-03

CONDITIONS: Multiple Myeloma; Quality of Life
Keywords: Multiple Myeloma; Quality of Life; Response Shift; Clinically Important Difference
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to determine Clinically important difference and Response shift in quality of life in patients with Multiple Myeloma.

DETAILED DESCRIPTION:
Multiple myeloma is a plasma cell tumor with an annual incidence of 6 pr. 100 000. In the absence of curative treatment, the aim of the therapy is not only to induce an objective response and a prolongation of survival but also to improve the patients quality of life.

This project will raise two problems which make QoL-data hard to interpret

1. In a clinical trial where many patients are included, statistically significant differences are obtained. However, there is widespread agreement that p-values do not indicate whether a particular finding has clinical significance because statistical significance does not necessarily equate to a meaningful difference or change in QoL. A crucial task for clinicians in interpreting trial-based QoL results is to determine if the observed change is clinically important to the patient.
2. When measuring changes in QoL in a pretest-posttest design,response shift can affect results. Patients with advanced disease can report surprisingly good QoL.Including response shift into quality of life research would allow a better understanding of changes in the QoL that patients report.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Myeloma
* Age > 18 years
* Informed consent

Exclusion Criteria:

* Terminal illness with life expectancy less than 3 months
* Unable to fill in a questionnaire in norwegian

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Multiple Myeloma in all fases in the south and east of Norway
Sampling Method: Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2006-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Finn Wisløff, MD, PhD, Principal Investigator — Ullevål University Hospital, Norway
Locations (1):
- Ullevaal University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Kvam AK, Wisloff F, Fayers PM. Minimal important differences and response shift in health-related quality of life; a longitudinal study in patients with multiple myeloma. Health Qual Life Outcomes. 2010 Aug 3;8:79. doi: 10.1186/1477-7525-8-79. PMID 20678240